CLINICAL TRIAL: NCT03345485
Title: A Phase 1/2 Study to Investigate the Safety, Pharmacokinetics and Efficacy of EDO-S101, a First-in-Class Alkylating Histone Deacetylase Inhibition (HDACi) Fusion Molecule, in Patients With Advanced Solid Tumors. Sub-study to Characterize the Effects of Tinostamustine at a Dose of 60mg/m2 Administered During a 60 Minutes Infusion on Cardiac Repolarization, in Patients With Advanced Solid Tumors. Sub-study to Characterize the Effects of Tinostamustine at a Dose of 80mg/m2 Administered During a 80 Minutes Infusion on Cardiac Repolarization, in Patients With Advanced Solid Tumors.
Brief Title: Study of the Safety, Pharmacokinetics and Efficacy of Tinostamustine in Patients With Advanced Solid Tumors.
Acronym: EDO-S101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EDO-S101-1002; 2020-004246-11 (EudraCT Number)
Record Dates: First submitted 2017-10-24; First posted 2017-11-17 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-06

CONDITIONS: Small Cell Lung Cancer; Soft Tissue Sarcoma; Triple-negative Breast Cancer; Ovarian Cancer; Endometrial Cancer
Keywords: Phase 1 (P1); Solid Tumor; Small Cell Lung Cancer (SCLC); Breast Cancer; Ovarian Cancer (OC); Soft Tissue Sarcoma (STS); Relapsed/Refractory; Triple Negative; Gastrointestinal stromal tumors (GIST); Epithelial cancer; Peritoneal cancer; Fallopian tube cancer; Metastatic; Advanced; Endometrial Cancer (EC); Phase 2 (P2); Corrected QT interval (QTc); System Organ Class (SOC); Preferred Term (PT); Day 1 (D1); Day 15 (D15); Treatment-Emergent Adverse Events (TEAEs); Investigational Medicinal Product (IMP); Polymorphonuclear cell (PMN); Progressive Response (PR); Stable disease (SD); Maximum administered dose (MAD); Dose-limiting toxicity (DLT)
MeSH Terms: conditions — Small Cell Lung Carcinoma; Sarcoma; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Breast Neoplasms; Recurrence; Gastrointestinal Stromal Tumors; Fallopian Tube Neoplasms; Neoplasm Metastasis | interventions — tinostamustine

STUDY DESIGN:
Intervention Model Description: In phase 1 (dose escalation phase) of the study, subjects were allocated sequentially.
  In phase 2, subjects were allocated in parallel to the various arms (cohorts) based on their cancer specifics.
  In the substudies 1 and 2, subjects were allocated into a single group in each substudy.
  Overall, the study model is described as Sequential as the study proceeded in phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 min) cohort 1 (Experimental)
  Interventions: Drug: Tinostamustine 60mg/m2 over 30min
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 min) cohort 2 (Experimental)
  Interventions: Drug: Tinostamustine 80mg/m2 over 30min
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 min) cohort 3 (Experimental)
  Interventions: Drug: Tinostamustine 100mg/m2 over 30min
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 min) cohort 4 (Experimental)
  Interventions: Drug: Tinostamustine 60mg/m2 over 60min
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 min) cohort 5 (Experimental)
  Interventions: Drug: Tinostamustine 80mg/m2 over 60min
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 min) cohort 6 (Experimental)
  Interventions: Drug: Tinostamustine 100mg/m2 over 60min
- Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Small Cell Lung Cancer (SCLC) cohort (Experimental)
  Interventions: Drug: Tinostamustine 80mg/m2 over 60min
- Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Soft Tissue Sarcoma (STS) cohort (Experimental)
  Interventions: Drug: Tinostamustine 80mg/m2 over 60min
- Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Triple Negative breast Cancer (TNBC) cohort (Experimental)
  Interventions: Drug: Tinostamustine 80mg/m2 over 60min
- Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Ovarian Cancer (OC) cohort (Experimental)
  Interventions: Drug: Tinostamustine 80mg/m2 over 60min
- Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Endometrial Cancer (EC) cohort (Experimental)
  Interventions: Drug: Tinostamustine 80mg/m2 over 60min
- Tinostamustine (EDO-S101) - Sub study 1 (SS1) (Experimental)
  Interventions: Drug: Tinostamustine 60mg/m2 over 60min
- Tinostamustine (EDO-S101) - Sub study 2 (SS2) (Experimental)
  Interventions: Drug: Tinostamustine 80mg/m2 over 80min

INTERVENTIONS:
Drug: Tinostamustine 60mg/m2 over 30min — Tinostamustine as a single agent was administered at doses of 60mg/m2 by intravenous infusion over 30 minutes on Days (D) 1 and 15 of each 28-day cycle.
  Other Names: EDO-S101
  Arms: Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 min) cohort 1
Drug: Tinostamustine 80mg/m2 over 30min — Tinostamustine as a single agent was administered at doses of 80mg/m2 by intravenous infusion over 30 minutes on Days (D) 1 and 15 of each 28-day cycle.
  Other Names: EDO-S101
  Arms: Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 min) cohort 2
Drug: Tinostamustine 100mg/m2 over 30min — Tinostamustine as a single agent was administered at doses of 100mg/m2 by intravenous infusion over 30 minutes on Days (D) 1 and 15 of each 28-day cycle.
  Other Names: EDO-S101
  Arms: Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 min) cohort 3
Drug: Tinostamustine 60mg/m2 over 60min — Tinostamustine as a single agent was administered at doses of 60mg/m2 by intravenous infusion over 60 minutes on Days (D) 1 and 15 of each 28-day cycle.
  Other Names: EDO-S101
  Arms: Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 min) cohort 4; Tinostamustine (EDO-S101) - Sub study 1 (SS1)
Drug: Tinostamustine 80mg/m2 over 60min — Tinostamustine as a single agent was administered at doses of 80mg/m2 by intravenous infusion over 60 minutes on Days (D) 1 and 15 of each 28-day cycle.
  Other Names: EDO-S101.
  Arms: Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 min) cohort 5; Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Endometrial Cancer (EC) cohort; Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Ovarian Cancer (OC) cohort; Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Small Cell Lung Cancer (SCLC) cohort; Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Soft Tissue Sarcoma (STS) cohort; Tinostamustine (EDO-S101) - Phase 2 Relapsed/refractory Triple Negative breast Cancer (TNBC) cohort
Drug: Tinostamustine 100mg/m2 over 60min — Tinostamustine as a single agent was administered at doses of 100mg/m2 by intravenous infusion over 60 minutes on Days (D) 1 and 15 of each 28-day cycle.
  Other Names: EDO-S101
  Arms: Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 min) cohort 6
Drug: Tinostamustine 80mg/m2 over 80min — Tinostamustine as a single agent was administered at doses of 80mg/m2 by intravenous infusion over 80 minutes on Days (D) 1 and 15 of each 28-day cycle.
  Other Names: EDO-S101
  Arms: Tinostamustine (EDO-S101) - Sub study 2 (SS2)

SUMMARY:
Tinostamustine (EDO-S101) is a first-in-class alkylating deacetylase inhibitor designed to improve drug access to deoxyribonucleic acid (DNA) strands, induce DNA damage and counteract its repair in cancer cells. The main purpose of this study is to assess the safety, tolerability and efficacy of Tinostamustine in subjects with advanced solid tumours. Subjects will be given Tinostamustine via intravenous infusion on Days 1 and 15 of a 4-week cycle, the dose and infusion time will vary depending on the phase of the study.

DETAILED DESCRIPTION:
The study consists of 2 phases and 2 sub-studies:

This study is a multi-centre, open-label phase 1/2 study of single agent EDO-S101 in subjects with advanced solid tumours.

Phase 1 part of the study is designed to determine the safety, tolerability, maximum tolerated dose (MTD), recommended phase 2 dose (RP2D) and the Pharmacokinetic (PK) of EDO-S101 as a single agent in patients with solid tumours who have progressed after at least one (1) line of therapy and for whom no other standard therapy with proven clinical benefit is available.

Phase 2 part of the study is designed to evaluate the overall response rate (ORR) of the RP2D, plus the rate of patients with stable disease (SD) at 4 or 6 months, depending on the type of solid tumour. The RP2D was determined after phase 1 to be 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and Day 15 of each 4-week treatment cycle.

In addition, two sub-studies are designed to better characterize the effect of EDO-S101: one at a dose of 60 mg/m2 administered over 60 minutes and the second at a dose of 80 mg/m2 administered over 80 minutes on cardiac repolarization (QTc) and other ECG parameters in the subjects with solid tumours.

Subjects were eligible for these studies if they had a histologically confirmed solid tumour, signed informed consent and met the inclusion/exclusion criteria. After providing informed consent, subjects were screened, and all procedures were performed as per protocol.

ELIGIBILITY:
Inclusion and exclusion criteria were reviewed for each potential patient during Screening. All eligible patients were treated with Tinostamustine employing sequential enrollment (i.e. as they qualify for participation). In the first phase of the trial (Phase 1), the dose received for each eligible patient was dependent on the requirements of the dose escalation scheme at the time the patient was enrolled. In the second phase of the trial (Phase 2), all patients were treated with the Tinostamustine at 80 mg/m2 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.

General Inclusion Criteria for Phase 1 and Phase 2 portions of Study:

1. Patient willing and able to sign the informed consent.
2. Patients age ≥18 years at signing the informed consent.
3. Life expectancy > 3 months.
4. Histologically confirmed diagnosis of advanced or metastatic solid tumors, disease should have progressed following at least one line of therapy and no other standard therapy with proven clinical benefit is available or recommended based on the investigator's individual risk-benefit assessment for the patient.
5. Patients with secondary metastasis to the central nervous system (CNS) are eligible if they have had brain metastases resected or have received radiation therapy ending at least 4 weeks prior to trial day 1 and they meet all of the following criteria:

   1. Residual neurological symptoms ≤Grade 1.
   2. No glucocorticoids requirement or patients may be receiving low doses of glucocorticoids providing the dose has been stable for at least 2 weeks prior to starting the trial medication.
   3. Follow-up imaging studies show no progression of treated lesions and no new lesions.
6. Evaluable disease; measurable on imaging as assessed by RECIST version 1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
8. Absolute neutrophil count (ANC) (polymorphonuclear cells [PMN] plus bands) >1,000/ μL.
9. Platelets ≥100,000 μL. Platelet transfusions within the 14 days before Day 1 of Cycle 1 is prohibited.
10. Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤ 3 upper limit of normal (ULN). In cases with liver involvement ALT/ AST ≤ 5× ULN.
11. Total bilirubin ≤1.5 mg/dL unless elevated due to known Gilbert's syndrome.
12. Creatinine ≤1.5 ULN.
13. Serum potassium and magnesium at least at the lowest limit of normal (LLN), before every IMP administration. If it is below the LLN, supplementation is permissible.
14. Female study participants of child-bearing potential and their partners, and male study participants who intend to be sexually active with a woman of child-bearing potential, must be willing to use at least two (2) highly effective forms of contraception. This should start from the time of study enrollment and continue throughout IMP administration. For female study participants of child-bearing potential this must continue using contraception for at least six (6) months after the last administration of the IMP. Female study participants should be willing to have a pregnancy test performed at screening, ≤ 1 day prior to day 1 of each IMP administration and at study treatment discontinuation. Male study participants who are sexually active with a woman of child-bearing potential should also use a condom during treatment and for at least ninety (90) days after the last administration of IMP. Vasectomized males are considered fertile; therefore, vasectomized partners and patients must be willing to use a secondary method of effective birth control. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient.

Exclusion Criteria Phase 1 and Phase 2 portions of Study:

To be eligible to participate in the trial, a patient cannot meet any of the following exclusion criteria:

1. Patients with primary central nervous system (CNS) cancer.
2. Patients with QTc interval (Fridericia's formula) >450 msec.
3. Patients who are on treatment with drugs known to prolong the QT/QTc interval.
4. Patients who are being treated with Valproic Acid for any of its indication (epilepsy, mood disorder).
5. Any serious medical condition that interferes with adherence to trial procedures.
6. Prior history of solid tumor malignancy diagnosed within the last three (3) years of study enrollment excluding adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer, in situ breast cancer, in situ prostate cancer (patients must have shown no evidence of active disease for 2 years prior to enrollment)
7. Pregnant or breast feeding females.
8. New York Heart Association (NYHA) stage III/IV congestive heart failure, arrhythmias not adequately controlled, or other significant co-morbidities [e.g. active infection requiring systemic therapy, history of human immunodeficiency virus (HIV) infection, or active Hepatitis B or Hepatitis C].
9. Use of other investigational agents within 28 days prior to the first dose of study drug, provided the patient has recovered from any related toxicities ≥Grade 1.
10. Steroid treatment within seven (7) days prior to trial treatment. Patients that require intermittent use of bronchodilators, topical steroids or local steroid injections will not be excluded from the study. Patients who have been stabilized to 10 mg Prednisolone orally (PO) once daily (QD) (or equivalent), daily (or less) at least seven (7) days prior to IMP administration are allowed.

Phase 2:

Patients must meet the cohort-specific inclusion/exclusion criteria in addition to the general inclusion/exclusion criteria for Phase 1 and Phase 2 study listed above.

Cohort 1: Relapsed/Refractory small cell lung cancer (SCLC)

1. Histologically or cytologically confirmed limited or extensive disease stage of SCLC.
2. Must have received at least 1 line of prior combination chemotherapy or biological therapy and no other standard therapy with proven clinical benefit is available or recommended based on the investigator's individual risk-benefit assessment for the patient.
3. At least 28 days should have elapsed since prior treatment as long as the patient has recovered from any related toxicities to ≤ Grade 1 (or ≤ Grade 2 for any symptomatic neuropathy or endocrinopathies).
4. Prior radiotherapy is acceptable provided the patient has recovered from any radiotherapy related acute toxicities.
5. The disease should be progressing during or relapsing after the previous treatment.
6. Presence of measurable disease as defined by RECIST version 1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion.

Cohort 2: Relapsed/Refractory Soft Tissue Sarcoma (STS)

1. Histologically confirmed diagnosis of advanced, unresectable, or metastatic soft tissue sarcoma not amenable to curative treatment with surgery or radiotherapy excluding: neuroblastoma, GIST, embryonal rhabdomyosarcoma, Kaposi sarcoma, chondrosarcoma, osteosarcoma or Ewing's sarcoma.
2. Must have received at least one prior line prior line chemotherapy or biological therapy regimen and no other standard therapy with proven clinical benefit is available or recommended based on the investigator's individual risk-benefit assessment for the patient. At least twenty-eight (28) days should have elapsed since prior chemotherapy, as long as the patient recovered from any related toxicities to ≤ Grade 1 (or ≤Grade 2 for any symptomatic neuropathy or endocrinopathies).
3. The disease should be progressing during or relapsing after the previous treatment.
4. Presence of measurable disease as defined by RECIST version 1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion.

Cohort 3: Relapsed/Refractory Triple Negative Breast Cancer (TNBC)

1. Histologically or cytologically confirmed locally advanced or metastatic Triple Negative Breast Cancer. Proven human epidermal growth factor receptor 2 (HER2) negative by immunohistochemistry (INH) or in situ hybridization (ISH) per per American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) guidelines.
2. Must have received at least one (1) line of chemotherapy or biological therapy and no other standard therapy with proven clinical benefit was available or recommended based on the Investigator's individual risk-benefit assessment for the subject.
3. At least three (3) weeks should have elapsed since prior chemotherapy as long as the subject recovered from acute toxicity of previous therapies to ≤ Grade 1 (or ≤ Grade 2 for any symptomatic neuropathy or endocrinopathies).
4. Prior radiotherapy was acceptable provided it was administered at least four (4) weeks (two (2) weeks for palliative, limited field radiation therapy) prior to starting treatment on this study and the subject recovered from any radiotherapy related acute toxicities.
5. The disease had to be progressing during or relapsing after the previous treatment.
6. Presence of measurable disease as defined by RECIST version 1.1. Tumour lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, were usually not considered measurable unless there had been demonstrated progression in the lesion.

Cohort 4: Patient Population: Relapsed/Refractory Ovarian Cancer (OC)

1. Histologically or cytologically confirmed advanced ovarian cancer: epithelial ovarian cancer, including primary peritoneal cancer or fallopian tube cancer (excluding borderline ovarian cancer, MMMT) of high grade serous histology, or high grade endometrioid cancer, that is resistant or refractory to platinum therapy and no other standard therapy with proven clinical benefit is available or recommended based on the investigator's individual risk-benefit assessment for the patient. Clear cell carcinomas are excluded. Patients with primary platinum refractory disease (failure to respond to initial platinum treatment or relapse within four (4) weeks) and patients with primary platinum resistant disease (progression within six (6) months of completing first line platinum-based therapy) are excluded from the study.
2. At least twenty eight (28) days should have elapsed since prior chemotherapy as long as the patient recovered from acute toxicity of previous therapies to ≤ Grade 1 (or ≤ Grade 2 for any symptomatic neuropathy or endocrinopathies).
3. The disease should be progressing during or relapsing after the previous treatment.
4. Presence of measurable disease as defined by RECIST version 1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion.

Cohort 5: Relapsed/Refractory Endometrial Cancer (EC)

1. Histologically or cytologically confirmed locally advanced or metastatic endometrial cancer (excluding leiomyosarcoma and carcinosarcoma)
2. Must have received at least one (1) line of chemotherapy and no other standard therapy with proven clinical benefit is available or recommended based on the investigator's individual risk-benefit assessment for the patient. At least three (3) weeks should have elapsed since prior chemotherapy or 5 half-lives, whichever is shorter, as long as the patient recovered from acute toxicity of previous therapies to ≤ Grade 1 (or ≤ Grade 2 for any symptomatic neuropathy or endocrinopathies).
3. Prior radiotherapy is acceptable provided it was administered at least four(4) weeks (two (2) weeks for palliative, limited field radiation therapy) prior to starting treatment on this trial and recovered from any radiotherapy related acute toxicities.
4. The disease should be progressing/relapsed during or after the previous treatment.
5. Presence of measurable disease as defined by RECIST version 1.1. Tumour lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, were usually not considered measurable unless there had been demonstrated progression in the lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2023-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, MD, Principal Investigator — Oregon Health and Science University; Ana Oaknin, MD, Principal Investigator — Head of Gynaecologic Cancer Program, Vall d'Hebron Institute of Oncology, Hospital Universitari Vall d'Hebron
Locations (13):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - University of Michigan, Ann Arbor, Michigan
  - New York University, New York, New York
  - Mary Crowley Cancer Research, Dallas, Texas
- Canada (3):
  - Juravinski Cancer Centre, Hamilton, Ontario, on
  - McGill University, Montreal, Quebec
  - BC Cancer-Vancouver, Vancouver, Vancouver, BC
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
- Erasmus MC Kanker Instituut, Rotterdam, Netherlands
- Spain (2):
  - Hospital Universitario La Paz, Madrid, Fuencarral-El Pardo
  - Hospital Universitari Vall d'Hebron, Barcelona, Horta-Guinardó

IPD SHARING:
Plan to Share IPD: Yes
Relevant patient listing data of de-identified patients may be reviewed
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available on request through Enquiries@napp.co.uk
Access Criteria: Available on request through Enquiries@napp.co.uk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by physicians at the study sites between Nov-2017 and Aug-2022.
Pre-assignment Details: Adults with histologically confirmed diagnosis of advanced or metastatic solid tumors, disease should have progressed during or following at least 1 previous line of therapy and no other standard therapy with proven clinical benefit is available or recommended based on the investigator's individual risk-benefit assessment for the patient.
Groups:
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min). Cohort 1: This is dose level 1 of the dose escalation phase (Phase 1) of the study.
  Tinostamustine at dose of 60mg/m2 administered i.v. over 30min on D1 and D15 of each 4-week cycle.
  The decision to escalate to the next dose level occurred after all 3 subjects completed the Dose-limiting toxicity (DLT) observation time and were evaluated for safety and toxicity.
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min). Cohort 2: This is dose level 2 of the dose escalation phase (Phase 1) of the study.
  Tinostamustine at dose of 80mg/m2 administered i.v. over 30min on D1 and D15 of each 4-week cycle.
  The decision to escalate to the next dose level occurred after all 3 subjects completed the Dose-limiting toxicity (DLT) observation time and were evaluated for safety and toxicity.
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min). Cohort 3.: This is dose level 3 of the dose escalation phase (Phase 1) of the study.
  Tinostamustine at dose of 100mg/m2 administered i.v. over 30min on D1 and D15 of each 4-week cycle.
  In the 30-minute infusion study drug dosing had to be delayed in subsequent cycles due to thrombocytopenia, which was associated with an extremely high Cmax of Tinostamustine. To ensure that subjects continue the study treatment safely, the Sponsor decided to stop the investigation of the 30-minute infusion time and open cohorts with the 60-minute infusion in 3 subjects with relapse/refractory solid tumors.
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min). Cohort 4: This is dose level 4 of the dose escalation phase (Phase 1) of the study.
  Tinostamustine at dose of 60mg/m2 administered i.v. over 60min on D1 and D15 of each 4-week cycle.
  The decision to escalate to the next dose level occurred after all 3 subjects completed the Dose-limiting toxicity (DLT) observation time and were evaluated for safety and toxicity.
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min). Cohort 5: This is dose level 5 of the dose escalation phase (Phase 1) of the study. Tinostamustine at dose of 80mg/m2 administered i.v. over 60min on D1 and D15 of each 4-week cycle.
  The decision to escalate to the next dose level occurred after all 3 subjects completed the Dose-limiting toxicity (DLT) observation time and were evaluated for safety and toxicity.
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min). Cohort 6: This is dose level 6 of the dose escalation phase (Phase 1) of the study.
  DLT of electrocardiogram QTc prolongation occurred 1 patient. Considering the DLT observed in this cohort and the rapid occurrence of treatment-induced thrombocytopenia (not meeting the DLT definitions), the SRC concluded as follows:
  * The dose of 100 mg/m2 was determined the MAD.
  * The dose level of 80 mg/m2 given i.v. over 60 minutes was determined to be the MTD
  * The dose level of 80 mg/m2 given i.v. over 60 minutes on Day 1 and Day 15 of each 4-week treatment cycle was determined to be the RP2D.
- Tinostamustine (EDO-S101) - Phase 2 SCLC Cohort.; Tinostamustine (EDO-S101) - Phase 2 STS Cohort.; Tinostamustine (EDO-S101) - Phase 2 TNBC Cohort.; Tinostamustine (EDO-S101) - Phase 2 OC Cohort.; Tinostamustine (EDO-S101) - Phase 2 EC Cohort.: Tinostamustine at dose of 80mg/m2 administered i.v. over 60min on D1 and D15 of each 4-week cycle.
- Tinostamustine (EDO-S101) - Substudy 1: Tinostamustine at dose of 60mg/m2 administered i.v. over 60min on D1 and D15 of each 4-week cycle.
- Tinostamustine (EDO-S101) - Substudy 2: Tinostamustine at dose of 80mg/m2 administered i.v. over 80min on D1 and D15 of each 4-week cycle.
Period: Overall Study
Arm/Group | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min). Cohort 1 | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min). Cohort 2 | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min). Cohort 3. | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min). Cohort 4 | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min). Cohort 5 | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min). Cohort 6 | Tinostamustine (EDO-S101) - Phase 2 SCLC Cohort. | Tinostamustine (EDO-S101) - Phase 2 STS Cohort. | Tinostamustine (EDO-S101) - Phase 2 TNBC Cohort. | Tinostamustine (EDO-S101) - Phase 2 OC Cohort. | Tinostamustine (EDO-S101) - Phase 2 EC Cohort. | Tinostamustine (EDO-S101) - Substudy 1 | Tinostamustine (EDO-S101) - Substudy 2
Started (Patients Treated) | 3 | 3 | 3 | 3 | 8 | 2 | 4 | 10 | 4 | 12 | 6 | 6 | 7
Completed (Phase 1: Patients are reported as completed if they have completed cycle 1. Phase 2: Patients who have at least 1 post-baseline tumour response assessment is reported as completed.) | 3 | 3 | 3 | 3 | 8 | 2 | 3 | 8 | 4 | 12 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 3 | 3
Not completed — Do not have a post-dose tumour assessment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics are summarised for Safety Population. Demographic information included age, sex, ethnicity, race, height, weight and BMI. Demographics and baseline characteristics were summarised descriptively. Subject demographics (sex, ethnicity, race, and age category) were presented using discrete summary statistics. Age, height, weight and BMI were presented using continuous summary statistics.
Groups:
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min). Cohort 1: Safety Population (All patients who received at least one (1) dose of study treatment at 60mg/m2 over a 30 minutes infusion time)
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min). Cohort 2: Safety Population (All patients who received at least one (1) dose of study treatment at 80mg/m2 over a 30 minutes infusion time)
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min). Cohort 3: Safety Population (All patients who received at least one (1) dose of study treatment at 100mg/m2 over a 30 minutes infusion time)
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min). Cohort 4: Safety Population (All patients who received at least one (1) dose of study treatment at 60mg/m2 over a 60 minutes infusion time)
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min). Cohort 5: Safety Population (All patients who received at least one (1) dose of study treatment at 80mg/m2 over a 60 minutes infusion time)
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min). Cohort 6: Safety Population (All patients who received at least one (1) dose of study treatment at 100mg/m2 over a 60 minutes infusion time)
- Tinostamustine (EDO-S101) - Phase 2 SCLC: Safety population (All patients who received at least one (1) dose of study treatment at 80mg/m2 over a 60 minutes infusion time) in patients with relapsed/refractory small cell lung cancer.
- Tinostamustine (EDO-S101) - Phase 2 STS: Safety population (All patients who received at least one (1) dose of study treatment at 80mg/m2 over a 60 minutes infusion time) in patients with relapsed/refractory soft tissue sarcoma.
- Tinostamustine (EDO-S101) - Phase 2 TNBC: Safety population (All patients who received at least one (1) dose of study treatment at 80mg/m2 over a 60 minutes infusion time) in patients with relapsed/refractory triple-negative breast cancer.
- Tinostamustine (EDO-S101) - Phase 2 OC: Safety population (All patients who received at least one (1) dose of study treatment at 80mg/m2 over a 60 minutes infusion time) in patients with relapsed/refractory ovarian cancer.
- Tinostamustine (EDO-S101) - Phase 2 EC: Safety population (All patients who received at least one (1) dose of study treatment at 80mg/m2 over a 60 minutes infusion time) in patients with relapsed/refractory endometrial cancer.
- Tinostamustine (EDO-S101) - Sub Study 1 (SS1): Subgroup treated with a dose of study treatment at 60 mg/m2 over 60 minutes infusion time.
- Tinostamustine (EDO-S101) - Sub Study 2 (SS2): Subgroup treated with a dose of study treatment at 80 mg/m2 over 80 minutes infusion time.
- Total: Total of all reporting groups
Arm/Group | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min). Cohort 1 | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min). Cohort 2 | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min). Cohort 3 | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min). Cohort 4 | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min). Cohort 5 | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min). Cohort 6 | Tinostamustine (EDO-S101) - Phase 2 SCLC | Tinostamustine (EDO-S101) - Phase 2 STS | Tinostamustine (EDO-S101) - Phase 2 TNBC | Tinostamustine (EDO-S101) - Phase 2 OC | Tinostamustine (EDO-S101) - Phase 2 EC | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 8 | 2 | 4 | 10 | 4 | 12 | 6 | 6 | 7 | 71
Age, Customized [Count of Participants; unit: Participants] — Age categories are defined per statistical analysis plan (SAP) document:
  1. < 65 years
  2. ≥ 65 or < 75 years
  3. ≥ 75 years
  Participants
    < 65 | 1 | 1 | 2 | 3 | 4 | 2 | 2 | 8 | 2 | 8 | 3 | 6 | 6 | 48
    ≥ 65 or < 75 | 2 | 2 | 1 | 0 | 4 | 0 | 2 | 2 | 1 | 3 | 3 | 0 | 0 | 20
    ≥ 75 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Age, Customized [Mean (Standard Deviation); unit: years] | 61.0 (12.12) | 60.7 (16.20) | 61.3 (8.74) | 54.0 (7.55) | 61.3 (13.55) | 56.5 (9.19) | 62.5 (6.56) | 53.2 (12.51) | 62.8 (18.39) | 61.6 (9.00) | 62.0 (8.74) | 49.5 (9.67) | 50.6 (17.18) | 57.87 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 4 | 2 | 2 | 6 | 4 | 12 | 6 | 5 | 4 | 52
  Male | 1 | 2 | 1 | 1 | 4 | 0 | 2 | 4 | 0 | 0 | 0 | 1 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 2 | 3 | 3 | 1 | 7 | 2 | 4 | 7 | 4 | 12 | 6 | 4 | 7 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  White | 3 | 2 | 1 | 3 | 6 | 2 | 4 | 8 | 3 | 10 | 4 | 5 | 6 | 57
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 4 | 0 | 0 | 0 | 7
  United States | 3 | 3 | 3 | 3 | 8 | 2 | 0 | 9 | 4 | 4 | 6 | 6 | 7 | 58
  Italy | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 5
  Spain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: Centimeters] — Height at Screening Population: During screening visit height was recorded for 69 patients
  Centimeters
    number analyzed (Participants) | 2 | 3 | 2 | 3 | 8 | 2 | 4 | 10 | 4 | 12 | 6 | 6 | 7 | 69
    (all) | 166.6 (12.87) | 173.6 (8.59) | 165.5 (24.75) | 162.3 (13.60) | 169.7 (16.13) | 164.8 (6.01) | 166.6 (12.98) | 166.3 (7.16) | 159.1 (6.78) | 160.3 (6.42) | 160.4 (3.57) | 165.4 (11.38) | 169.5 (10.55) | 165.07 (10.30)
Weight [Mean (Standard Deviation); unit: Kilograms] — Weight at Screening Population: During screening visit weight was recorded for 70 patients
  Kilograms
    number analyzed (Participants) | 3 | 3 | 2 | 3 | 8 | 2 | 4 | 10 | 4 | 12 | 6 | 6 | 7 | 70
    (all) | 74.2 (27.82) | 92.5 (7.51) | 75.3 (11.74) | 93.7 (8.87) | 71.2 (22.68) | 87.6 (25.31) | 72.7 (38.14) | 78.6 (29.17) | 62.4 (16.30) | 68.4 (15.23) | 66.1 (13.94) | 97.9 (27.79) | 74.7 (17.16) | 76.16 (22.65)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI (Body Mass Index) at screening Population: During screening visit BMI was recorded for 69 patients
  kg/m^2
    number analyzed (Participants) | 2 | 3 | 2 | 3 | 8 | 2 | 4 | 10 | 4 | 12 | 6 | 6 | 7 | 69
    (all) | 31.620 (1.7819) | 30.850 (3.9493) | 27.775 (3.9810) | 35.970 (6.1309) | 24.539 (6.5699) | 32.675 (11.7026) | 25.148 (8.6313) | 28.206 (9.9631) | 24.483 (4.9410) | 26.616 (5.7605) | 25.677 (5.2798) | 36.168 (11.1967) | 26.200 (6.8562) | 28.048 (7.7735)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE V4.03 on Phase 1
Description: All TEAEs was reported from the first dose of study drug through the time of study drug discontinuation (at any time or Day 28 of the last treatment Cycle). All treatment-related TEAEs was followed until resolution or stabilization. For the purpose of regulatory reporting requirements, causal relationships of definite, probable, and possible was considered treatment-related.
  Number of patients experiencing treatment-related adverse events (TEAE) as assessed by CTCAE v4.03. (June 2010).
Time Frame: From each patient's time of first dose administration to discontinuation of study drug (at any time or D28 of the last treatment cycle), up to 6 months.
Population: The safety analysis summarised TEAEs for all treated subjects using discrete summaries at the subject and event level by system organ class (SOC) and preferred term (PT). Treatment-related TEAEs were summarised similarly. TEAEs were also summarised by the grade of National Cancer Institute Common Terminology Criteria for Adverse Events. All AEs were coded using the MedDRA® version 24.0
Measure: Count of Participants; unit: Participants
Groups:
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min) Cohort 1: Patients who received Tinostamustine at 60mg/m2 (30min) on D1 and D15 of a 4-week cycle
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min) Cohort 2: Patients who received Tinostamustine at 80mg/m2 (30min) on D1 and D15 of a 4-week cycle
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min) Cohort 3: Patients who received Tinostamustine at 100mg/m2 (30min) on D1 and D15 of a 4-week cycle
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min) Cohort 4: Patients who received Tinostamustine at 60mg/m2 (60min) on D1 and D15 of a 4-week cycle
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min) Cohort 5: Patients who received Tinostamustine at 80mg/m2 (60min) on D1 and D15 of a 4-week cycle
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min) Cohort 6: Patients who received Tinostamustine at 100mg/m2 (60min) on D1 and D15 of a 4-week cycle
Arm/Group | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min) Cohort 1 | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min) Cohort 2 | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min) Cohort 3 | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min) Cohort 4 | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min) Cohort 5 | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min) Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 8 | 2
Participants
  Investigations | 3 | 3 | 3 | 3 | 6 | 2
  Gastrointestinal disorders | 3 | 3 | 2 | 1 | 8 | 2
  Blood and lymphatic system disorders | 1 | 3 | 2 | 3 | 4 | 1
  General disorders and administration site conditions | 1 | 2 | 2 | 2 | 5 | 1
  Nervous system disorders | 1 | 1 | 2 | 1 | 3 | 2
  Skin and subcutaneous tissue disorders | 1 | 2 | 1 | 1 | 2 | 0
  Metabolism and nutrition disorders | 1 | 0 | 0 | 1 | 3 | 1
  Injury, poisoning and procedural complications | 0 | 1 | 0 | 0 | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 0 | 0 | 1 | 0 | 1 | 0
  Cardiac disorders | 0 | 0 | 0 | 0 | 1 | 0
  Musculoskeletal and connective tissue disorders | 0 | 0 | 0 | 0 | 1 | 0
  Vascular disorders | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Clinical Benefit Response Rate in Selected Solid Tumor Cohorts on Phase 2
Description: The Clinical Benefit Response Rate is calculated as the number of patients with Clinical Benefit Response divided by number of patients in the FAS (in the respective cohort). Clinical Benefit Response is defined as patients achieving stable disease with a duration of at least 12 weeks (84 days).
  Summary subjects analysed were 36.
Time Frame: From start treatment and assessed after every 2 cycles until determination of stable disease and follow up for up to 84 days.
Population: All subjects who received at least 1 dose of study treatment were included in the Full Analysis (FA) Population. Efficacy analyses were performed on data from all subjects in the FA Population
Measure: Number (90% Confidence Interval); unit: percentage of patients
Groups:
- Tinostamustine (EDO-S101) - Phase 2 SCLC: A dose of study treatment at 80 mg/m2 administered over 1 hour in patients with relapsed/refractory small cell lung cancer.
- Tinostamustine (EDO-S101) - Phase 2 STS: A dose of study treatment at 80 mg/m2 administered over 1 hour in in patients with relapsed/refractory soft tissue sarcoma.
- Tinostamustine (EDO-S101) - Phase 2 TNBC: A dose of study treatment at 80 mg/m2 administered over 1 hour in patients with relapsed/refractory Triple-negative breast cancer.
- Tinostamustine (EDO-S101) - Phase 2 OC: A dose of study treatment at 80 mg/m2 administered over 1 hour in patients with relapsed/refractory Ovarian Cancer.
- Tinostamustine (EDO-S101) - Phase 2 EC: A dose of study treatment at 80 mg/m2 administered over 1 hour in patients with relapsed/refractory Endometrial Cancer.
Arm/Group | Tinostamustine (EDO-S101) - Phase 2 SCLC | Tinostamustine (EDO-S101) - Phase 2 STS | Tinostamustine (EDO-S101) - Phase 2 TNBC | Tinostamustine (EDO-S101) - Phase 2 OC | Tinostamustine (EDO-S101) - Phase 2 EC
Number analyzed (Participants) | 4 | 10 | 4 | 12 | 6
percentage of patients | 0 [0 to 52.7] | 40.0 [15.0 to 69.6] | 50.0 [9.8 to 90.2] | 50.0 [24.5 to 75.5] | 50.0 [15.3 to 84.7]

3. Primary Outcome: Highest Change From Baseline in QTcF in Sub-studies
Description: QTcF: corrected QT interval [QTc] using Fridericia's formula) and other electrocardiogram (ECG) parameters in subjects with solid tumours who have progressed after at least 1 line of therapy and for whom no other standard therapy with proven clinical benefit is available.
  Within each cycle a Change from baseline (CfB) is calculated for QTcF relative to the baseline value of day 1 of the cycle. QTcF CfB= QTcF Post-dose value - QTcF pre-dose value of D1 ECG Parameters: 4-hours ECG holter monitoring in C1 and ECGs during EDO-S101 administration.
  Continuous variables the mean and standard deviation are presented together with the total number of observations and the number of missing and non-missing values.
Time Frame: From cycle 1 and at every cycle on treatment days D1 and D15, assessed pre-dose and post-start of infusion at 30 and 80mins (Substudy 2 - up to 6 months) and 30, 60, 90, 120 and 180mins (substudy 1 - up to 6 months).
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Tinostamustine (EDO-S101) - Sub Study 1 (SS1): 6 Patients treated with 60 mg/m2 as a single agent of Tinostamustine administered over 60 minutes infusion time
- Tinostamustine (EDO-S101) - Sub Study 2 (SS2): 7 Patients treated with 80 mg/m2 as a single agent of Tinostamustine administered over 80 minutes infusion time
Arm/Group | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2)
Number analyzed (Participants) | 6 | 7
msec | 53.33 (23.777) | 33.24 (12.588)

4. Secondary Outcome: Treatment-related Adverse Events on Phase 2 and Sub Studies
Description: Number of patients experiencing treatment-related adverse events (TEAE) as assessed by CTCAE v4.03, June 2010, with the exception that assessment of QTc prolongations constituting adverse events (AEs) of special interest were based on NCI CTCAE version 5.0, November 2017.
  All subjects who received at least 1 dose of study treatment were included in the Safety Population. Safety analyses were performed on data from all subjects in the Safety Population.
  Adverse events are reported on a patient basis. The percentages are calculated using the number of patients in the Safety Analysis Set as the denominator.
Time Frame: From each patient's time of informed consent to discontinuation of study drug (at any time or D28 of the last treatment cycle), up to 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Tinostamustine (EDO-S101) - Phase 2 SCLC Cohort: Patients with Relapsed/refractory small cell lung cancer (SCLC)
- Tinostamustine (EDO-S101) - Phase 2 STS Cohort: Patients with Relapsed/refractory soft tissue sarcoma (STS)
- Tinostamustine (EDO-S101) - Phase 2 TNBC Cohort: Patients with Relapsed/refractory triple-negative breast cancer (TNBC)
- Tinostamustine (EDO-S101) - Phase 2 OC Cohort: Patients with Relapsed/refractory Ovarian Cancer (OC)
- Tinostamustine (EDO-S101) - Phase 2 EC Cohort: Patients with Relapsed/refractory Endometrial Cancer (EC)
- Tinostamustine (EDO-S101) - Sub Study 1 (SS1): Subgroup treated with a dose of 60 mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Sub Study 2 (SS2): Subgroup treated with a dose of 80 mg/m2 over 80 minutes infusion time of EDO-S101
Arm/Group | Tinostamustine (EDO-S101) - Phase 2 SCLC Cohort | Tinostamustine (EDO-S101) - Phase 2 STS Cohort | Tinostamustine (EDO-S101) - Phase 2 TNBC Cohort | Tinostamustine (EDO-S101) - Phase 2 OC Cohort | Tinostamustine (EDO-S101) - Phase 2 EC Cohort | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2)
Number analyzed (Participants) | 4 | 10 | 4 | 12 | 6 | 6 | 7
Participants
  Gastrointestinal disorders | 2 | 4 | 3 | 12 | 4 | 2 | 2
  Investigations | 3 | 3 | 2 | 8 | 5 | 3 | 2
  Blood and lymphatic system disorders | 2 | 4 | 2 | 7 | 3 | 3 | 3
  General disorders and administration site conditions | 2 | 3 | 1 | 9 | 5 | 2 | 1
  Metabolism and nutrition disorders | 1 | 1 | 1 | 4 | 3 | 1 | 0
  Nervous system disorders | 2 | 2 | 0 | 3 | 3 | 1 | 0
  Skin and subcutaneous tissue disorders | 1 | 3 | 0 | 4 | 1 | 0 | 0
  Musculoskeletal and connective tissue disorders | 1 | 1 | 0 | 1 | 0 | 1 | 1
  Respiratory, thoracic and mediastinal disorders | 1 | 1 | 1 | 0 | 1 | 1 | 0
  Vascular disorders | 0 | 2 | 0 | 2 | 1 | 0 | 0
  Cardiac disorders | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Injury, poisoning and procedural complications | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Infections and infestations | 0 | 1 | 0 | 0 | 0 | 0 | 2

5. Secondary Outcome: Progression Free Survival (PFS) Time for Phase 2 and Sub Studies
Description: PFS was defined as the number of days between the date of the first dose of treatment of a patient and the first date of disease progression, start of a subsequent anti-cancer therapy, or death of the patient.
Time Frame: From patient's first dose until first documented progression/start of subsequent anti-cancer therapy/death from any cause, whichever came first, up to 26 months.
Measure: Median (90% Confidence Interval); unit: days
Groups:
- Tinostamustine (EDO-S101) - Phase 2 SCLC Cohort: Progression-free survival (PFS) time for patients with small cell lung cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Phase 2 STS Cohort: Progression-free survival (PFS) time for patients with soft tissue sarcoma who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Phase 2 TNBC Cohort: Progression-free survival (PFS) time for patients with triple-negative breast cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Phase 2 OC Cohort: Progression-free survival (PFS) time for patients with ovarian cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Phase 2 EC Cohort: Progression-free survival (PFS) time for patients with endometrial cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Sub Study 1 (SS1): Progression-free survival (PFS) time for patients with solid tumour who received 60 mg/m2 of EDO-S101 administered over 1 hour
- Tinostamustine (EDO-S101) - Sub Study 2 (SS2): Progression-free survival (PFS) time for patients with solid tumour who received 80 mg/m2 of EDO-S101 administered over 80 minutes
Arm/Group | Tinostamustine (EDO-S101) - Phase 2 SCLC Cohort | Tinostamustine (EDO-S101) - Phase 2 STS Cohort | Tinostamustine (EDO-S101) - Phase 2 TNBC Cohort | Tinostamustine (EDO-S101) - Phase 2 OC Cohort | Tinostamustine (EDO-S101) - Phase 2 EC Cohort | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2)
Number analyzed (Participants) | 4 | 10 | 4 | 12 | 6 | 6 | 7
days | 54.0 [50.0 to NA] — Could not be calculated due to insufficient number of participants with events | 56.0 [50.0 to 236.0] | 85.0 [58.0 to NA] — Could not be calculated due to insufficient number of participants with events | 63.0 [44.0 to 97.0] | 87.0 [33.0 to 107.0] | 177.0 [62.0 to NA] — Could not be calculated due to insufficient number of participants with events | 65.0 [23.0 to NA] — Could not be calculated due to insufficient number of participants with events

6. Secondary Outcome: Overall Survival (OS) Time for Phase 2 and Sub Studies
Description: Overall survival is defined as the number days between the date of the first dose of treatment and the date of death. If no date of death is recorded the Overall Survival time is censored at the Last available visit date.
  Phase 2: To determine the overall survival (OS) time for subjects with solid tumours.
  SS1:To determine the overall survival (OS) time for subjects who received 60 mg/m2 of EDO-S101 during a 60-minute Infusion.
  SS2: To determine the overall survival (OS) time for subjects who received 80 mg/m2 of EDO-S101 during a 80-minute Infusion.
Time Frame: From patient's first dose until first documented progression/start of subsequent anti-cancer therapy/death from any cause, whichever came first, up to 42 months.
Population: Full Analysis Set (FAS): All patients who received at least 1 dose of trial treatment and had at least 1 post-baseline response evaluation.
Measure: Median (90% Confidence Interval); unit: Days
Groups:
- Tinostamustine (EDO-S101) - Phase 2 SCLC Cohort: Overall survival (OS) time for patients with small cell lung cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Phase 2 STS Cohort: Overall survival (OS) time for patients with soft tissue sarcoma who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Phase 2 TNBC Cohort: Overall survival (OS) time for patients with triple-negative breast cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Phase 2 OC Cohort: Overall survival (OS) time for patients with ovarian cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Phase 2 EC Cohort: Overall survival (OS) time for patients with endometrial cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour on Day 1 and 15 of each 4-week treatment cycle.
- Tinostamustine (EDO-S101) - Sub Study 1 (SS1): Overall survival (OS) time for patients with solid tumour who received 60 mg/m2 of EDO-S101 administered over 1 hour.
- Tinostamustine (EDO-S101) - Sub Study 2 (SS2): Overall survival (OS) time for patients with solid tumour who received 80 mg/m2 of EDO-S101 administered over 80 minutes.
Arm/Group | Tinostamustine (EDO-S101) - Phase 2 SCLC Cohort | Tinostamustine (EDO-S101) - Phase 2 STS Cohort | Tinostamustine (EDO-S101) - Phase 2 TNBC Cohort | Tinostamustine (EDO-S101) - Phase 2 OC Cohort | Tinostamustine (EDO-S101) - Phase 2 EC Cohort | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2)
Number analyzed (Participants) | 4 | 10 | 4 | 12 | 6 | 6 | 7
Days | 114.5 [85.0 to NA] — Could not be calculated due to insufficient number of participants with events | 346.5 [76.0 to NA] — Could not be calculated due to insufficient number of participants with events | 218.5 [58.0 to NA] — Could not be calculated due to insufficient number of participants with events | 261.0 [121.0 to NA] — Could not be calculated due to insufficient number of participants with events | 127.0 [33.0 to NA] — Could not be calculated due to insufficient number of participants with events | 177.0 [62.0 to NA] — Could not be calculated due to insufficient number of participants with events | 139.0 [23.0 to NA] — Could not be calculated due to insufficient number of participants with events

7. Secondary Outcome: Maximum Duration of Response (DoR) Time for Phase 2 and Sub Studies
Description: The duration of objective response is measured from the date of the first tumor response assessment with an Investigator's Overall Response of CR or PR (whichever status is recorded first) until the date of progression or death. DoR is presented by subject.
Time Frame: From patient's first overall response of CR or PR, until disease progression/subsequent anti-cancer therapy/death from any cause, up to 24 months.
Population: Number of participants is zero in some of the arms as no participants achieved a response of CR or PR.
Measure: Number; unit: days
Groups:
- Tinostamustine (EDO-S101) - Phase 2 STS Cohort: Duration of response for patients with soft tissue sarcoma cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour.
- Tinostamustine (EDO-S101) - Phase 2 OC Cohort: Duration of response for patients with ovarian cancer who received 80 mg/m2 of EDO-S101 administered over 1 hour.
- Tinostamustine (EDO-S101) - Sub Study 1 (SS1): Duration of response for patients with solid tumour who received 60 mg/m2 of EDO-S101 administered over 1 hour.
Arm/Group | Tinostamustine (EDO-S101) - Phase 2 STS Cohort | Tinostamustine (EDO-S101) - Phase 2 OC Cohort | Tinostamustine (EDO-S101) - Sub Study 1 (SS1)
Number analyzed (Participants) | 1 | 1 | 1
days | 51 | 52 | 734

8. Secondary Outcome: Objective Response Rate (ORR) and the Clinical Benefit Rate (CBR) That Persists for at Least Four (4) Months in Selected Solid Tumor Cohorts on Sub Studies
Description: To determine the objective response rate (ORR) and the clinical benefit rate (CBR [Complete Response (CR), Partial Response (PR) plus durable Stable Disease (SD)]) in Sub Studies.
  SD was regarded as durable if, after observing SD, the first observation of PD was at least 84 days after the start of study treatment.
Time Frame: From start of treatment, assessed every 2 cycles, until first documented complete CR, PR or SD, up to 6 months. If SD, assessment continued every 2 cycles until CR/PR/death (up to 6 months)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Tinostamustine (EDO-S101) - Sub Study 1 (SS1): To determine the objective response rate (ORR) (complete response [CR] plus partial response [PR]) of any duration, plus the rate of subjects with stable disease (SD) of at least 12-week duration at a dose of 60 mg/m2 administered over 1 hour.
- Tinostamustine (EDO-S101) - Sub Study 2 (SS2): To determine the objective response rate (ORR) (complete response [CR] plus partial response [PR]) of any duration, plus the rate of subjects with stable disease (SD) of at least 12-week duration at a dose of 80 mg/m2 administered over 80 minutes.
Arm/Group | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2)
Number analyzed (Participants) | 6 | 7
percentage of participants
  Objective Response Rate (CR+PR) (%) | 16.7 [0.9 to 58.2] | 0 [0 to 34.8]
  Clinical Benefit Response Rate (CR+PR+durable SD) % | 50.0 [15.3 to 84.7] | 14.3 [0.7 to 52.1]

9. Secondary Outcome: Number of Participants With Duration of Stable Disease (SD) That Persists for at Least 4 Months in Selected Solid Tumor Cohorts in Sub Studies.
Description: Duration of SD, was defined as the number of days between the date of the first dose of treatment and the first date of disease progression or death.
  SD was regarded as durable if, after observing SD, the first observation of progression disease was at least 84 days after the start of study treatment.
Time Frame: as for outcome 8
Population: Analysis population includes only those subjects who achieved stable disease (SD). The Duration of SD (was regarded as durable if, after observing SD, the first observation of PD was at least 84 days after the start of study treatment) was based of number of patients with Best Overall Stable Disease Response.
Measure: Count of Participants; unit: Participants
Groups:
- Tinostamustine (EDO-S101) - Sub Study 1 (SS1): A dose of 60 mg/m2 administered over 60 minutes on D1 and D15 of 4-week cycles
- Tinostamustine (EDO-S101) - Sub Study 2 (SS2): A dose of 80 mg/m2 administered over 80 minutes on D1 and D15 of 4-week cycles.
Arm/Group | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2)
Number analyzed (Participants) | 2 | 1
Participants
  <84 days | 0 | 0
  ≥84 days | 2 | 1

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) in Phase 2 and Sub Studies
Time Frame: Blood samples were collected over a period of 24hr (phase 2 and sub-study 1) and 30hr (sub-study 2) on Cycle 1 Day 1 and Day 15.
Population: All enrolled subjects in the Safety Population with at least 1 quantifiable pre-dose and 1 quantifiable post-dose PK plasma concentration in Cycle 1 were included in the PK Population. PK analyses were performed using the PK population. 48 subjects of the Safety Population were included in the PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram(s)/millilitre
Groups:
- Phase 2 All Cohorts: A dose of 80 mg/m2 administered over 60 minutes on D1 and D15 of 4-week cycles.
Arm/Group | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2) | Phase 2 All Cohorts
Number analyzed (Participants) | 6 | 7 | 35
nanogram(s)/millilitre
  EDO-S101 concentration, Cycle 1 D1 | 1150 (15.8) | 1210 (11.3) | 1620 (43.3)
  EDO-S101 concentration, Cycle 1 D15: number analyzed (Participants) | 5 | 6 | 34
  EDO-S101 concentration, Cycle 1 D15 | 999 (38.6) | 1040 (21.2) | 1540 (41.5)
  M2 metabolite concentration, Cycle 1 D1: number analyzed (Participants) | 5 | 5 | 24
  M2 metabolite concentration, Cycle 1 D1 | 2.18 (65.4) | 2.32 (65.5) | 1.92 (77.9)
  M2 metabolite concentration, Cycle 1 D15: number analyzed (Participants) | 3 | 1 | 24
  M2 metabolite concentration, Cycle 1 D15 | 2.31 (105) | 2.91 (NA) — Not calculated due to insufficient data | 1.98 (63.3)
  M8 metabolite concentration, Cycle 1 D1 | 37.4 (17.0) | 27.0 (36.5) | 47.7 (50.2)
  M8 metabolite concentration, Cycle 1 D15: number analyzed (Participants) | 5 | 6 | 34
  M8 metabolite concentration, Cycle 1 D15 | 31.2 (46.3) | 24.6 (33.3) | 49.8 (43.7)

11. Secondary Outcome: Area Under the Curve [AUC(0-t)] in Phase 2 and Sub Studies.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2) | Phase 2 All Cohorts
Number analyzed (Participants) | 6 | 7 | 35
ng.h/mL
  EDO-S101 concentration, Cycle 1 D1 | 938 (41.9) | 1680 (22.6) | 1490 (40.9)
  EDO-S101 concentration, Cycle 1 D15: number analyzed (Participants) | 5 | 6 | 34
  EDO-S101 concentration, Cycle 1 D15 | 943 (53.7) | 1390 (28.7) | 1520 (41.7)
  M2 metabolite concentration, Cycle 1 D1: number analyzed (Participants) | 5 | 5 | 24
  M2 metabolite concentration, Cycle 1 D1 | 5.19 (420) | 12.4 (1430) | 0.865 (248)
  M2 metabolite concentration, Cycle 1 D15: number analyzed (Participants) | 3 | 1 | 24
  M2 metabolite concentration, Cycle 1 D15 | 2.32 (9060) | 48.6 (NA) — Not calculated due to insufficient data | 1.32 (163)
  M8 metabolite concentration, Cycle 1 D1 | 36.0 (80.5) | 54.4 (61.2) | 47.7 (48.3)
  M8 metabolite concentration, Cycle 1 D15: number analyzed (Participants) | 5 | 6 | 34
  M8 metabolite concentration, Cycle 1 D15 | 40.9 (94.1) | 35.2 (33.7) | 53.3 (44.8)

12. Secondary Outcome: Summary of Tmax in in Phase 2 and Sub Studies.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2) | Phase 2 All Cohorts
Number analyzed (Participants) | 6 | 7 | 35
hours
  EDO-S101 concentration, Cycle 1 D1 | 0.750 [0.250 to 0.750] | 1 [0.750 to 1.33] | 0.750 [0.250 to 1.25]
  EDO-S101 concentration, Cycle 1 D15: number analyzed (Participants) | 5 | 6 | 35
  EDO-S101 concentration, Cycle 1 D15 | 0.750 [0.5 to 0.750] | 0.875 [0.167 to 1.33] | 0.750 [0 to 1.25]
  M2 metabolite concentration, Cycle 1 D1: number analyzed (Participants) | 5 | 5 | 35
  M2 metabolite concentration, Cycle 1 D1 | 1 [0.250 to 6] | 1.58 [0.750 to 24] | 1.00 [0.25 to 2.00]
  M2 metabolite concentration, Cycle 1 D15: number analyzed (Participants) | 3 | 1 | 35
  M2 metabolite concentration, Cycle 1 D15 | 1 [0.250 to 24] | 3.50 [3.50 to 3.50] | 1.00 [0 to 6]
  M8 metabolite concentration, Cycle 1 D1 | 0.750 [0.250 to 1] | 1 [1 to 1.33] | 0.750 [0.250 to 1.50]
  M8 metabolite concentration, Cycle 1 D15: number analyzed (Participants) | 5 | 6 | 35
  M8 metabolite concentration, Cycle 1 D15 | 0.750 [0.500 to 0.750] | 1.33 [1 to 1.33] | 0.750 [0 to 1.25]

13. Secondary Outcome: Clearance of Tinostamustine and Metabolites in Phase 2 and Substudies
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/m^2
Arm/Group | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2) | Phase 2 All Cohorts
Number analyzed (Participants) | 6 | 7 | 35
mL/h/m^2
  EDO-S101 concentration, Cycle 1 D1: number analyzed (Participants) | 4 | 3 | 28
  EDO-S101 concentration, Cycle 1 D1 | 69800 (48.7) | 56000 (23.9) | 50800 (41.1)
  EDO-S101 concentration, Cycle 1 D15: number analyzed (Participants) | 3 | 2 | 21
  EDO-S101 concentration, Cycle 1 D15 | 89600 (19.5) | 49600 (58.3) | 53600 (45.2)
  M2 metabolite concentration, Cycle 1 D1 | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived. | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived. | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived.
  M2 metabolite concentration, Cycle 1 D15 | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived. | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived. | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived.
  M8 metabolite concentration, Cycle 1 D1: number analyzed (Participants) | 3 | 3 | 35
  M8 metabolite concentration, Cycle 1 D1 | 2410000 (54.2) | 2270000 (22.4) | NA (NA) — M8 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived.
  M8 metabolite concentration, Cycle 1 D15: number analyzed (Participants) | 2 | 3 | 35
  M8 metabolite concentration, Cycle 1 D15 | 1240000 (14.8) | 1740000 (40.8) | NA (NA) — M8 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived.

14. Secondary Outcome: Summary of Half-life of Tinostamustine in Phase 2 and Substudies.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Tinostamustine (EDO-S101) - Sub Study 1 (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2) | Phase 2 All Cohorts
Number analyzed (Participants) | 6 | 7 | 35
hour
  EDO-S101 concentration, Cycle 1 D1: number analyzed (Participants) | 4 | 3 | 28
  EDO-S101 concentration, Cycle 1 D1 | 0.919 (38) | 2.14 (185) | 0.70 (54)
  EDO-S101 concentration, Cycle 1 D15: number analyzed (Participants) | 3 | 2 | 20
  EDO-S101 concentration, Cycle 1 D15 | 0.678 (45.8) | 4.03 (2150) | 0.704 (51.2)
  M2 metabolite concentration, Cycle 1 D1 | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived. | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived. | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived.
  M2 metabolite concentration, Cycle 1 D15 | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived. | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived. | NA (NA) — M2 metabolite plasma concentrations were either below the limit of quantification, or a regression line could not be fitted to calculate elimination rate constant due to R square value not meeting acceptance criteria. Therefore clearance could not be derived.
  M8 metabolite concentration, Cycle 1 D1: number analyzed (Participants) | 3 | 7 | 17
  M8 metabolite concentration, Cycle 1 D1 | 0.602 (30.2) | 1.22 (96.8) | 0.414 (49)
  M8 metabolite concentration, Cycle 1 D15: number analyzed (Participants) | 3 | 7 | 7
  M8 metabolite concentration, Cycle 1 D15 | 2.30 (153) | 2.48 (99.7) | 4.43 (553)

ADVERSE EVENTS:
Time Frame: Phase (P) 1: From time of first dose to study drug discontinuation (at any time or Day 28 of the last treatment cycle), followed up to stabilisation/resolution (up to 33 months). P2 and Substudies (SS): From point of ICF signature to study drug discontinuation (at any time or Day 28 of the last treatment cycle), followed up to stabilisation or resolution (P2 and SS1 -up to 49 months) or (SS2 up to 18 months).
Description: TEAE will be captured from the first day of study drug dosing through discontinuation of study drug (at any time or Day 28 of the last treatment cycle). Serious adverse events (SAEs) will be reported from first day of study drug until 30 days after last treatment.
  P1: All AEs were coded using the MedDRA® version 24.0 and P2 using the MedDRA® version 20.0.
Groups:
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min) Cohort 1: Patients who received 60mg/m2 over 30 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min) Cohort 2: Patients who received 80mg/m2 over 30 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min) Cohort 3: Patients who received 100mg/m2 over 30 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min) Cohort 4; Tinostamustine (EDO-S101) - Sub Study (SS1): Patients who received 60mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min) Cohort 5: Patients who received who 80mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min) Cohort 6: Patients who received who 100mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 2 SCLC: Patient with relapsed/refractory SCLC who received 80mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 2 STS: Patient with relapsed/refractory STS who received 80mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 2 TNBC: Patient with relapsed/refractory TNBC who received 80mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 2 OC: Patient with relapsed/refractory OC who received 80mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Phase 2 EC: Patient with relapsed/refractory EC who received 80mg/m2 over 60 minutes infusion time of EDO-S101
- Tinostamustine (EDO-S101) - Sub Study 2 (SS2): Patients who received 80mg/m2 over 80 minutes infusion time of EDO-S101
Arm/Group | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min) Cohort 1 | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min) Cohort 2 | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min) Cohort 3 | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min) Cohort 4 | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min) Cohort 5 | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min) Cohort 6 | Tinostamustine (EDO-S101) - Phase 2 SCLC | Tinostamustine (EDO-S101) - Phase 2 STS | Tinostamustine (EDO-S101) - Phase 2 TNBC | Tinostamustine (EDO-S101) - Phase 2 OC | Tinostamustine (EDO-S101) - Phase 2 EC | Tinostamustine (EDO-S101) - Sub Study (SS1) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/3 | 2/8 | 0/2 | 1/4 | 3/10 | 2/4 | 2/12 | 3/6 | 4/6 | 2/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 2/3 | 3/3 | 5/8 | 2/2 | 0/4 | 6/10 | 1/4 | 7/12 | 4/6 | 6/6 | 0/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 8/8 | 2/2 | 4/4 | 10/10 | 4/4 | 12/12 | 6/6 | 6/6 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min) Cohort 1 (N=3) | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min) Cohort 2 (N=3) | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min) Cohort 3 (N=3) | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min) Cohort 4 (N=3) | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min) Cohort 5 (N=8) | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min) Cohort 6 (N=2) | Tinostamustine (EDO-S101) - Phase 2 SCLC (N=4) | Tinostamustine (EDO-S101) - Phase 2 STS (N=10) | Tinostamustine (EDO-S101) - Phase 2 TNBC (N=4) | Tinostamustine (EDO-S101) - Phase 2 OC (N=12) | Tinostamustine (EDO-S101) - Phase 2 EC (N=6) | Tinostamustine (EDO-S101) - Sub Study (SS1) (N=6) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2) (N=7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (30 Min) Cohort 1 (N=3) | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (30 Min) Cohort 2 (N=3) | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (30 Min) Cohort 3 (N=3) | Tinostamustine (EDO-S101) - Phase 1 - 60mg/m2 (60 Min) Cohort 4 (N=3) | Tinostamustine (EDO-S101) - Phase 1 - 80mg/m2 (60 Min) Cohort 5 (N=8) | Tinostamustine (EDO-S101) - Phase 1 - 100mg/m2 (60 Min) Cohort 6 (N=2) | Tinostamustine (EDO-S101) - Phase 2 SCLC (N=4) | Tinostamustine (EDO-S101) - Phase 2 STS (N=10) | Tinostamustine (EDO-S101) - Phase 2 TNBC (N=4) | Tinostamustine (EDO-S101) - Phase 2 OC (N=12) | Tinostamustine (EDO-S101) - Phase 2 EC (N=6) | Tinostamustine (EDO-S101) - Sub Study (SS1) (N=6) | Tinostamustine (EDO-S101) - Sub Study 2 (SS2) (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 3 (7) | 3 (6) | 3 (16) | 3 (6) | 1 (1) | 1 (1) | 2 (4) | 2 (3) | 5 (7) | 4 (15) | 2 (6) | 0 (0)
Cyclic neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (8) | 1 (1) | 2 (2) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 3 (4) | 2 (3) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Catheter site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (4) | 2 (2) | 2 (4) | 6 (14) | 1 (1) | 1 (2) | 4 (5) | 1 (2) | 3 (6) | 5 (8) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (5) | 1 (3) | 0 (0) | 1 (2) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 4 (4) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (3) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 1 (1) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anticipatory anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: EDO-S101-1002 Phase 2 protocol v8.1 (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT03345485/Prot_000.pdf
  • Study Protocol: EDO-S101-1002 Substudy 2 (80/80) protocol v6.7 (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03345485/Prot_001.pdf
  • Study Protocol: EDO-S101-1002 Substudy 1 (60/60) protocol v6.2 (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03345485/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03345485/SAP_004.pdf